CLINICAL TRIAL: NCT06870292
Title: Assessment of the Effectiveness and Safety of Posterior Nasal Nerve Combined with Anterior Ethmoid Neurotomy in Patients with Idiopathic Rhinitis: a Multicentre, Randomised, Parallel-controlled Study
Brief Title: Posterior Nasal Nerve Combined with Anterior Ethmoid Neurotomy for Idiopathic Rhinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Yu (Other)
Responsible Party: Sponsor-Investigator, Xu Yu, Dr., Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2024-K232; 2023YFC2507905 (Other Grant/Funding Number: National Key Research and Development Program of China)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Rhinitis
Keywords: Idiopathic Rhinitis; posterior nasal nerve neurotomy; anterior ethmoid neurotomy; surgical treatment; neuroimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Posterior nasal nerve combined with anterior ethmoid neurotomy group (Experimental): Subjects will undergo posterior nasal nerve combined with anterior ethmoid neurotomy under nasal endoscope.
  Interventions: Procedure: Posterior nasal nerve combined with anterior ethmoid neurotomy
- Drug therapy group (Active Comparator): Subjects will be treated with medication according to guideline recommendations when nasal symptoms such as nasal obstruction, rhinorrhea, itching, and sneezing occur. Oral antihistamines (Loratadine) or nasal antihistamines (Azelastine) are preferred, and nasal hormones (Budesonide), or a combination of two or three drugs, may be used in severe cases.
  Interventions: Drug: Drug therapy group

INTERVENTIONS:
Procedure: Posterior nasal nerve combined with anterior ethmoid neurotomy — First, a vertical incision was made in the posterior portion of the middle nasal turbinate. Dissection was performed along the bone to elevate the mucosal flap to expose the thick orbital process of the vertical plate of the palatine bone and the sphenopalatine foramen. The 3-4 mm of mucosal and submucosal neurovascular bundles surrounding the sphenopalatine foramen were subjected to full radiofrequency ablation, directly to the bone. The mucoperiosteal flap is reposited back. The bilateral nasal cavity was packed with Merocel nasal pack and hemostasis was achieved.
  The anterior ethmoidal nerves of the lateral nasal branch and septal branch of the nasal cavity were cut off with a plasma treatment needle. Below 30°, the mucous membrane of the posterior lateral wall of the nasal colliculus was cut down to the bone surface using the needle of the nasal endoscope plasma therapy instrument. The contralateral side was then treated in the same way, with an arc cut line and a length of 2cm.
  Arms: Posterior nasal nerve combined with anterior ethmoid neurotomy group
Drug: Drug therapy group — Subjects will be treated with medication according to guideline recommendations when nasal-related symptoms occur. Oral antihistamines or nasal antihistamines are preferred, and nasal hormones (budesonide nasal spray), or a combination of two or three drugs, may be used in severe cases.
  Arms: Drug therapy group

SUMMARY:
The present study was a randomised, parallel controlled, open-label, multicentre clinical study. The trial was divided into two groups, the posterior nasal nerve combined with anterior ethmoid neurotomy group (group A) and the conventional drug treatment group (group B). Patients with idiopathic rhinitis (IR) who met the inclusion criteria were included in a 7-day introductory period of nasal spray hormone (Budesonide nasal spray) treatment. Subjects with IR who met the randomization criteria after the introductory period were randomized 1:1 to either group A or group B for a 1-year treatment follow-up study. In group A, subjects will undergo the posterior nasal nerve combined with anterior ethmoid neurotomy. In group B, subjects will be treated with medication according to guideline recommendations when nasal-related symptoms occur. Oral antihistamines (Loratadine) or nasal antihistamines (Azelastine Hydrochloride) are preferred, and nasal hormones (Budesonide nasal spray), or a combination of two or three drugs, may be used in severe cases. Participants will be evaluated for safety and efficacy throughout the entire three-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients signed the free and informed consent form and understood the explanation of the study.
2. patients with IR between 18 and 65 years and their body mass index (BMI) should be ≥19 kg/m2 and ≤24 kg/m2.
3. Patients diagnosed with idiopathic rhinitis （IR）that were defined as nonsmoking patients with at least 2 nasal complaints of nasal obstruction, rhinorrhea, itching, and/or sneezing for more than 1 hour a day and for more than 1 year.
4. Patients with negative skin prick test (SPT) responses or sIgE
5. Nasal cytological exam with eosinophilia less than 20%.
6. Patients had a Total Nasal Symptom Score (TNSS) of ≥6 and a subscore of nasal discharge ≥2 and a subscore of nasal congestion ≥1.

Exclusion Criteria:

1. Patients with colored secretions, inflammation，nasal polyps, chronic sinusitis, nasal tumours.
2. Patients with other chronic rhinitis such as occupational rhinitis, drug rhinitis, gustatory rhinitis, hormonal rhinitis, atrophic rhinitis, etc.
3. Patients with anatomic nasal abnormalities responsible for nasal symptoms.
4. Patients with nasal/sinus surgery 3 months before the study.
5. Patients with severe mental illness.
6. Patients with uncontrolled asthma, systemic disorders or malignancies.
7. Patients with history of chronic smoking, substance abuse, drug use, and/or excessive alcohol consumption.
8. Patients in pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Combined symptom and medication score (CSMS) | 3rd postoperative months
  The combined symptom and medication score (CSMS) is a validated composite metric widely used in clinical research and practice to holistically assess the severity and control of rhinitis. It integrates both subjective symptom burden and objective medication use into a single quantitative score.A questionnaire was used to evaluate the CSMS.

SECONDARY OUTCOMES:
Combined symptom and medication score (CSMS) | 6th and 12th postoperative months
  The combined symptom and medication score (CSMS) is a validated composite metric widely used in clinical research and practice to holistically assess the severity and control of rhinitis. It integrates both subjective symptom burden and objective medication use into a single quantitative score.A questionnaire was used to evaluate the CSMS.
Total nasal symptoms score (TNSS) | 3rd, 6th, and 12th postoperative months
  The total nasal symptoms score (TNSS) is a patient-reported outcome tool widely utilized to quantify the severity of nasal symptoms in allergic rhinitis (AR) and other rhinologic conditions. It provides a standardized, composite assessment of key nasal symptoms including nasal congestion, rhinorrhea, sneezing, and nasal itching. A questionnaire was used to evaluate the TNSS.
Rhinoconjunctivitis quality of life questionnaire (RQLQ) | 3rd, 6th, and 12th postoperative months
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) is a validated, patient-reported outcome measure specifically designed to assess the impact of rhinoconjunctivitis on patients' daily functioning and overall well-being. It incluges 28 items grouped into 7 domains: nasal symptoms, ocular symptoms, practical problems, activity limitations, emotional impact, sleep disturbances, general health perceptions.
Rhinitis Control Assessment Test (RCAT) | 3rd, 6th, and 12th postoperative months
  The RCAT is a patient-reported assessment tool designed to evaluate the level of control over rhinitis symptoms, assisting clinicians in evaluating treatment efficacy and adjusting management strategies.It typically consists of six items assessing the frequency of symptoms (such as nasal congestion, rhinorrhea, and sneezing) and their impact on daily life over the past week. For the RCAT, an internationally recognized questionnaire was used for measurement.
Substance P（SP）、Vasoactive Intestinal Peptide（VIP）、Calcitonin Gene-Related Peptide（CGRP）、Neuropeptide Y（NPY） | 3rd, 6th, and 12th postoperative months
  Neuropeptide substance P (SP), vasoactive intestinal peptide (VIP), calcitonin gene-related peptide (CGRP) and neuropeptide Y (NPY) were measured in nasal secretions using ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu R, Dong L, Mao H, Wang J, Ma D, Sun J. Clinical study on the treatment of moderate to severe persistent allergic rhinitis by posterior nasal nerve combined with anterior ethmoid neurotomy. Pak J Med Sci. 2022 Sep-Oct;38(7):1888-1892. doi: 10.12669/pjms.38.7.5561. PMID 36246705
- [Background] Balai E, Gupta KK, Jolly K, Darr A. Posterior nasal nerve neurectomy for the treatment of rhinitis: a systematic review and meta-analysis. Eur Ann Allergy Clin Immunol. 2023 May;55(3):101-114. doi: 10.23822/EurAnnACI.1764-1489.268. Epub 2022 Sep 6. PMID 36066203
- [Background] Baroody FM, Gevaert P, Smith PK, Ziaie N, Bernstein JA. Nonallergic Rhinopathy: A Comprehensive Review of Classification, Diagnosis, and Treatment. J Allergy Clin Immunol Pract. 2024 Jun;12(6):1436-1447. doi: 10.1016/j.jaip.2024.03.009. Epub 2024 Mar 11. PMID 38467330
- [Background] Hellings PW, Klimek L, Cingi C, Agache I, Akdis C, Bachert C, Bousquet J, Demoly P, Gevaert P, Hox V, Hupin C, Kalogjera L, Manole F, Mosges R, Mullol J, Muluk NB, Muraro A, Papadopoulos N, Pawankar R, Rondon C, Rundenko M, Seys SF, Toskala E, Van Gerven L, Zhang L, Zhang N, Fokkens WJ. Non-allergic rhinitis: Position paper of the European Academy of Allergy and Clinical Immunology. Allergy. 2017 Nov;72(11):1657-1665. doi: 10.1111/all.13200. Epub 2017 Jun 2. PMID 28474799
- [Background] Lieberman PL, Smith P. Nonallergic Rhinitis: Treatment. Immunol Allergy Clin North Am. 2016 May;36(2):305-19. doi: 10.1016/j.iac.2015.12.007. Epub 2016 Feb 26. PMID 27083104